CLINICAL TRIAL: NCT03613974
Title: Successful Popliteal Block Using Lidocaine; What is the Minimum Effective Anesthesia Concentration (MEAC90)
Brief Title: Minimum Anaesthesia Concentration of Lidocaine Required for Sciatic Popliteal Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Healthpoint Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Muhammad Taha, Consultant of anesthesia, Healthpoint Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Healthpoint Hospital
Record Dates: First submitted 2018-07-20; First posted 2018-08-03 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Orthopedic Procedures
Keywords: foot and ankle; day case surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Masking Description: the patients and the assessment staff will not be aware with the given lidocaine concentration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lidocaine concentraion (Experimental): the popliteal block will be performed (once) in all patients using 20 ml of lidoacine. The response of a patient determined the lidocaine concentration given to the next patient (a biased-coin design up-down sequential method). If a patient had a negative response (failed block), the lidocaine concentration was increased by 0.1% w/v in the next patient. If a patient had a positive response (successful block), the next patient was randomized to receive the same lidocaine concentration (with probability of 0.89), or to receive a concentration 0.1% w/v less (with probability of 0.11).
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — patients will receive different lidocaine concentrations

SUMMARY:
using a biased-coin design up-down sequential method, different concentration of lidocaine will be used for popliteal block After 45 successful block (positive response), the data will be used to calculate the minimum lidocaine concentration that can result in successful popliteal block in 90% of patients

DETAILED DESCRIPTION:
The response of a patient determined the lidocaine concentration given to the next patient (a biased-coin design up-down sequential method). If a patient had a negative response, the lidocaine concentration was increased by 0.1% w/v in the next patient. If a patient had a positive response, the next patient was randomized to receive the same lidocaine concentration (with probability of 0.89), or to receive a concentration 0.1% w/v less (with probability of 0.11).

ELIGIBILITY:
Inclusion Criteria:

* orthopedic foot or ankle surgery
* day case surgery

Exclusion Criteria: patients

* <18y,
* ASA class greater >III,
* obese (BMI >30),
* patients with low body weight, who required lidocaine dose is of more than 4.5mg.kg-1
* peripheral neuropathy,
* motor weakness,
* infection at the injection site
* any contraindications for medications in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
successful popliteal block (positive response) | 30 min to 3 hour after the block
  Sensory block will be assessed using pinprick sensation. Complete sensory block = unable to recognize pinprick sensation. Intra-operative pain will be assessed using Visual Analogue Scale (VAS) 0 = No pain, 10 = Worst imaginable pain.
  Successful block = complete sensory block + pain free surgery (VAS = 0).

SECONDARY OUTCOMES:
motor block | 30 min after the block
  degree of motor weakness
motor recovery | 3 hours till full recovery
  complete recover of the motor power
analgesic duration | few hours after block
  requesting painkiller

IPD SHARING:
Plan to Share IPD: Undecided